CLINICAL TRIAL: NCT00004109
Title: A Phase I Study of Preoperative Concurrent Chemoradiation for High-Risk Extremity and Trunk Soft Tissue Sarcomas
Brief Title: Doxorubicin Plus External-Beam Radiation Therapy in Treating Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID97-335; P30CA016672 (NIH); MDA-ID-97335 (Other: UT MD Anderson Cancer Center); NCI-G99-1598; CDR0000067332 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-12-10; First posted 2004-03-15 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Sarcoma
Keywords: stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; Doxorubicin; External-Beam RT; XRT; cancer; PREOPERATIVE CONCURRENT CHEMORADIATION; EXTREMITY SOFT TISSUE SARCOMAS; TRUNK SOFT TISSUE SARCOMAS; Concurrent Chemoradiation; Surgical Resection; Localized Extremity Soft Tissue Sarcomas; Body Wall Soft Tissue Sarcomas
MeSH Terms: conditions — Sarcoma; Neoplasms | interventions — Doxorubicin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxorubicin + External-Beam RT (Experimental)
  Interventions: Drug: Doxorubicin Hydrochloride; Radiation: Radiation Therapy (RT)

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride — Doxorubicin dose will not exceed 20 mg/m2 per week IV over 4 days every week for 5 weeks
  Other Names: doxorubicin
Radiation: Radiation Therapy (RT) — External-beam radiotherapy at a dose of 50 Gy (2.0 x 25 fractions, weeks 1-5).
  Other Names: RT; Radialtherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of doxorubicin plus external-beam radiation therapy in treating patients who have soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity and maximum tolerated dose of doxorubicin when combined with external beam radiotherapy in patients with high risk soft tissue sarcomas of the extremity or trunk. II. Assess the radiographic and pathologic response rates to this preoperative regimen in the subset of these patients with measurable disease.

OUTLINE: This is a dose escalation study of doxorubicin. Patients receive doxorubicin intravenous (IV) bolus followed immediately by doxorubicin IV over 4 days every week for 5 weeks in the absence of unacceptable toxicity. Patients with measurable disease receive external beam radiotherapy 5 days a week for 5 weeks concurrently with doxorubicin treatment. Patients with measurable disease undergo surgical resection of the residual mass 4-7 weeks following completion of chemoradiation. Patients who have no measurable disease and have undergone prereferral excision undergo surgical resection of the prior surgical scar and tumor bed followed by external beam radiotherapy 5 days a week for 5 weeks. Cohorts of 3 patients receive escalating doses of doxorubicin until the maximum tolerated dose (MTD) is determined. Patients are followed every 3 months for 3 years, every 4 months for 2 years, and then annually for 5 years.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study at a rate of 5-6 patients per month.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have cytologic or histologic proof of large (>5 mc), Grade III, resectable soft tissue sarcoma of the extremity or trunk (AJCC Stage IIIB). Patients with The American Joint Committee on Cancer (AJCC) Stage IIB tumors (Grade II) greater than 8 cms will also be eligible.
2. Patients may have measurable or non-measurable disease (C/P pre-referral excision).
3. Patients may have had prior doxorubicin (up to a total doxorubicin dose of 450 mg/m2).
4. Patients may have a prior history of malignancy (at the discretion of the Principal Investigator).
5. Patients must have Karnofsky Point Scale (P.S.)> of >70 or Xubrod P.S. of 0 or 1.
6. Patients must have: Absolute neutrophil count (ANC) > 1,500 cells/mm; platelet count > 100,000 platelets/ml; serum creatinine <1.8 mg/dl, aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) < 3 times normal, total bilirubin < 1.5mg/dl; for patients with cumulative Adriamycin 450 mg/M2, EF >50%.
7. Women of childbearing potential must not be pregnant or breast feeding and must practice adequate contraception.

Exclusion Criteria:

1. Patients must not have had prior radiation therapy (XRT) in the area of the primary tumor, and the anticipated XRT field must not include the perineum, scrotum, or vaginal introitus.
2. Patients with uncontrolled coexisting medical conditions are excluded.
3. Patient must not be pregnant or brest feeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1998-03; Primary Completion 2001-09 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Continousouly during 5 weeks treatment
  MTD of doxorubicin intravenous (IV) based on presence of dose limiting toxicities. For dose-finding purposes, a dose-limiting toxicity (DLT) was defined as grade 3 or greater treatment-related cutaneous toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Peter W. Pisters, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org